CLINICAL TRIAL: NCT02649023
Title: Pre- and Early Postoperative Deep Venous Thrombosis in Patients Undergoing Oncological Hepatic or Panreatic Resection
Brief Title: Deep Venous Thrombosis After Hepatobiliopancreatic Surgery
Acronym: POPLITEA
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-05
Record Dates: First submitted 2015-12-07; First posted 2016-01-07 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Hepatectomy; Pancreatectomy
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Circulating tumor cells evaluation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Patients with deep venous thrombosis: All patients will be screened for deep venous thrombosis on postoperative day 3. Patients with a positive finding will be grouped in arm "A"
- B: Patients without deep venous thrombosis: All patients will be screened for deep venous thrombosis on postoperative day 3. Patients with a negative finding will be grouped in arm "B"

SUMMARY:
To investigate the incidence of pre- and early postoperative deep venous thrombosis in patients undergoing hepatobiliopancreatic surgery, as well as potential corresponding risk factors with special attention to circulating tumor cells.

DETAILED DESCRIPTION:
Thromboembolic events are a common cause of morbidity and mortality in oncological patients. Up to 20% of cancer patients suffer from venous thromboembolism (VTE) induced by the underlying malignancy itself. Oncologic gastrointestinal surgery is a well-known risk factor for VTE. About 4-6% of patients undergoing elective hepatobiliopanreatic surgery develop a deep venous thrombosis (DVT) or pulmonary embolism. However, there are no data referring to the incidence of DVT shortly ahead of the surgical event, implementing that a certain percentage of postoperative DVT might have already been acquired before the operation. Furthermore, most studies only evaluate the rate of symptomatic VTE. In this study, all patients undergoing hepatobiliopancreatic surgery will be screened for deep venous thrombosis the day before surgery, on the third postoperative day (primary endpoint) and 90 days after the operation with a 2-point compression sonography of the lower extremities. The development of a symptomatic VTE (DVT or pulmonary embolism) will be recorded as secondary endpoint. Risk factors, perioperative morbidity / mortality and presence of circulating tumor cells will be analyzed with regard to VTE incidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective oncological liver or pancreatic resection
* Age equal or greater than 18 years
* Written informed consent

Exclusion Criteria:

* Preexistent coagulopathy
* History of previous VTE
* benign disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective oncological liver or pancreatic resection
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Deep venous thrombosis on day 3 after surgery | 3 days
  Patients will be screened for deep venous thrombosis using a compression ultrasonography at the popliteal and common femoral vein. In case of a pathological finding, a complete compression duplex sonography of the lower extremities will be used for specification.

SECONDARY OUTCOMES:
Symptomatic deep venous thrombosis or pulmonary embolism during hospital stay | 30 days
  Patients who develop clinical signs of a DVT like swelling of the leg, pain or tenderness in the leg, increased warmth, red or discolored skin of the leg, will be diagnosed by complete compression duplex sonography for confirmation of a deep venous thrombosis. Patients who develop clinical signs of pulmonary embolism like unexplained shortness of breath, pain with deep breathing, coughing of blood, chest pain with electrocardiographic signs of right ventricular stress will be diagnosed by CT pulmonary angiography for confirmation of central or peripheral pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Nuh Rahbari, MD, Principal Investigator — Department of GI, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden
Locations (1):
- Department of GI, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No